CLINICAL TRIAL: NCT01952392
Title: Study on the Prevention of Cardiovascular Events by Antiplatelet Agents After Acute Coronary Syndrome
Brief Title: Prevention of Cardiovascular Events by Antiplatelet Agents After Acute Coronary Syndrome
Acronym: AReMIS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CFR-BRI-2012/1
Record Dates: First submitted 2013-08-21; First posted 2013-09-30 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Acute Coronary Syndrome
Keywords: Effectiveness study; Acute coronary Syndrome; Real-life; France
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Control group: Patients aged 18 years or more with an acute coronary syndrome, agreed to participate and able to answer an interview in French and/or providing the details of an alternative replier (proxy) if necessary
- Case group: Patients aged 18 years or more with a history of acute coronary syndrome (i.e. a recurrent MI after myocardial history or unstable angina), agreed to participate and able to answer an interview in French and/or providing the details of an alternative replier (proxy) if necessary

SUMMARY:
Prevention of cardiovascular events by antiplatelet agents after acute coronary syndrome

DETAILED DESCRIPTION:
AReMIS (Antiplatelet and Recurrent Myocardial Infarction Study) To compare the relative risk of new myocardial infarction (recurrent myocardial infarction or 'rMI') in patients with a history of acute coronary syndrome ('ACS': unstable angina or myocardial infarction), using ticagrelor, clopidogrel or prasugrel (if applicable) or none of these treatments, where aspirin is considered a covariate.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 years or more, both genders, with an acute coronary syndrome (ACS), agreed to participate and able to respond to an interview in French and/or providing the details of an alternative replier (proxy) if necessary.

No Exclusion Criteria.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or more, both genders,with an acute coronary syndrome, agreed to participate and able to respond to an interview in French and/or providing the details of an alternative replier (proxy) if necessary.
Sampling Method: Probability Sample
Enrollment: 4992 (Actual)
Dates: Start 2013-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Medical information | At baseline visit
  History of coagulation and vascular disorders History of cerebrovascular accidents Cardiovascular risk factors
Drug exposure | Current
  Current exposure: within 24 hours (before date of recurrent MI). Exposure to clopidogrel, ticagrelor, prasugrel, aspirin, other antiplatelet drugs.
Drug exposure | Recent
  Recent exposure: in the week (7 days) preceding the recurrent MI. Exposure to clopidogrel, ticagrelor, prasugrel, aspirin, other antiplatelet drugs.
Drug exposure | Past
  Past exposure: more than a week (7 days) before the recurrent MI and until the ACS index. Exposure to clopidogrel, ticagrelor, prasugrel, aspirin, other antiplatelet drugs.

SECONDARY OUTCOMES:
Other medical events of interest | During follow-up (up to 12 months)
  rMI, stroke, bleeding, death

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Paris, France

REFERENCES:
- See also: CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1819&filename=CSR_Synopsis_AReMIS.pdf